CLINICAL TRIAL: NCT02044406
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Oral Doses of BI 1181181 in Healthy Male Volunteers in a Partially Randomised, Single-blind, Placebo-controlled Trial, and Investigation of Relative Bioavailability and the Effect of Food on the Pharmacokinetics of BI 1181181(Open-label, Randomised, Three-way Cross-over Design)
Brief Title: Safety, Tolerability, Pharmacokinetics of Single Rising Oral Doses of BI 1181181 in Healthy Male Volunteers, Including Investigation of the Effect of Food on the Bioavailability of BI 1181181
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1344.1; 2013-002868-88 (EudraCT Number: EudraCT)
Record Dates: First submitted 2014-01-22; First posted 2014-01-24 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-10

CONDITIONS: Healthy

ARMS (2):
- 1 BI 1181181 single rising dose part (Experimental): single rising doses of BI 1181181
  Interventions: Drug: BI 1181181; Drug: Placebo to BI 1181181
- 2 BI 1181181 bioavailability part (Experimental): bioavailability, food effect part of BI 11881181
  Interventions: Drug: BI 1181181, R; Drug: BI 1181181, T2; Drug: BI 1181181, T1

INTERVENTIONS:
Drug: BI 1181181 — single dose (low to high dose)
  Arms: 1 BI 1181181 single rising dose part
Drug: BI 1181181, R — powder for oral solution
  Arms: 2 BI 1181181 bioavailability part
Drug: BI 1181181, T2 — tablet, fasted
  Arms: 2 BI 1181181 bioavailability part
Drug: Placebo to BI 1181181 — Placebo to BI 1181181
  Arms: 1 BI 1181181 single rising dose part
Drug: BI 1181181, T1 — tablet, fed
  Arms: 2 BI 1181181 bioavailability part

SUMMARY:
To investigate the safety, tolerability, pharmacokinetics (including dose proportionality assessment), and pharmacodynamics of single rising oral doses of BI 1181181 (Single rising dose (SRD) part) Secondly, to investigate the relative bioavailability of the tablet versus the powder for oral solution (PfOS) and the effect of food on the pharmacokinetics of BI 1181181 (Bioavailability/Food effect (BA/FE) part)

ELIGIBILITY:
Inclusion criteria:

* Healthy males according to the investigator's assessment, as based on the following criteria: a complete medical history including a physical examination, vital signs blood pressure (BP), pulse rate (PR), 12-lead ECG, and clinical laboratory tests
* Age 18 to 50 years (incl.)
* Body mass index (BMI) 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation

Exclusion criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and judged clinically relevant by the investigator
* Repeated measurement of systolic blood pressure < 90 mmHg and >= 140 mmHg at screening
* Repeated measurement of diastolic blood pressure < 55 and >= 90 mmHg at screening
* Repeated measurement of pulse rate < 50 bpm and > 90 bpm at screening
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2014-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Number (%) of subjects with drug-related adverse events (AEs) | up to 72 h
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point) | up to 72 h
Cmax (maximum measured concentration of the analyte in plasma) | up to 72 h

SECONDARY OUTCOMES:
Aet1-t2 (Amount of analyte that is eliminated in urine from the time point t1 to timepoint t2 after single dose administration) | up to 72 h
Cmax (maximum measured concentration of the analyte in plasma) | up to 72 h
tmax (time from dosing to maximum measured concentration of the analyte in plasma) | up to 72 h
AUC0-infinity (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 72 h
t1/2 (terminal half-life of the analyte in plasma) | up to 72 h

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1344.1.1 Boehringer Ingelheim Investigational Site, Ingelheim, Germany